CLINICAL TRIAL: NCT04977947
Title: Reducing Health Disparities Through an Adaptive Healthy Eating Program for Underserved Infants in a Home Visiting Program
Brief Title: Healthy Eating for My Infant (HEMI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Cathy Stough, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-0698
Record Dates: First submitted 2021-05-20; First posted 2021-07-27 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Obesity
Keywords: Obesity prevention; Behavioral intervention; Health disparities; Trauma informed; Child nutrition; Responsive feeding; Infant
MeSH Terms: conditions — Pediatric Obesity | interventions — Diet, Healthy

STUDY DESIGN:
Intervention Model Description: Infants will be assigned to either the treatment or control condition (standard care).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Eating for My Infant Intervention (Experimental): Participants and their parents will participate in a 6 session intervention targeting healthy introduction of complementary foods, and responsive feeding and mealtime behaviors. Intervention sessions will occur when the infant is 3, 4, 5, 6, 7, and 8 months of age.
  Interventions: Behavioral: Healthy Eating for My Infant
- Control (No Intervention): Participants and their parents will complete baseline and post-treatment study visits to assess study outcomes. They will receive no intervention.

INTERVENTIONS:
Behavioral: Healthy Eating for My Infant — The intervention targets problem solving to overcome barriers, behavioral rehearsal and practice of healthy behaviors, promoting readiness to change, goal setting, self-monitoring, and behavioral tracking. Two standard treatment modules will be provided to each family by a study interventionist focusing on infant nutritional requirements, responsive feeding, and mealtime behaviors. Two additional treatment modules will be selected to address the unique needs articulated by each family (e.g., food insecurity, eating healthy on a limited income, emotional eating, engaging other caregivers, maternal mental health). Modules will consider the influence of maternal trauma history and mental health on feeding and eating behavior. The intervention also includes two peer counselor-led sessions during which families can discuss implementation of recommendations and barriers to change with a member of their community who can problem solve and support change.
  Other Names: HEMI
  Arms: Healthy Eating for My Infant Intervention

SUMMARY:
Infants from underserved and minority backgrounds are at increased risk for obesity and poor feeding and nutrition outcomes, but obesity prevention programs tailored specifically to the needs of these infants are lacking. The current study takes a community-engaged approach to development and delivery of an adaptively tailored obesity prevention program delivered via home visiting to target infant eating and feeding (Healthy Eating for My Infant; HEMI).

DETAILED DESCRIPTION:
Poor dietary habits and obesity-risk begin early in infancy. Infants from underserved and minority backgrounds experience disparate rates of poor nutritional outcomes and subsequent health disparities related to obesity. Each infant and their family experiences a unique set of risk factors and barriers to healthy eating. However, obesity prevention programs that are culturally and contextually relevant for underserved families and adapted based on the needs of individual families are lacking. The current study will develop an obesity prevention program, Healthy Eating for My Infant (HEMI), using a community-engaged approach involving community members in development and delivery of the program. HEMI targets healthy infant feeding through six monthly sessions with infants 3-8 months old. The program will be delivered as a supplement to an already existing evidence-based home visiting program, Every Child Succeeds (ECS), serving families with primarily low income and ethnic/racial minority backgrounds.

Development of an adaptive and effective obesity prevention program meeting the needs of underserved infants is critical for addressing health disparities in infant eating and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Infant enrolled in the Every Child Succeeds (ECS) program
* Infant age is < 2 months at study recruitment
* Infant born at > 37 weeks gestation
* Infant is a singleton
* Maternal age is > 18 years (in order to consent for child to participate)
* Mother is fluent in English or Spanish

Exclusion Criteria:

* Infant has a major medical condition that requires specialized feeding

Ages: 2 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathleen Stough, PhD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Eating for My Infant Intervention | Control
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Eating for My Infant Intervention | Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: days] | 71.67 (9.42) | 73.53 (8.93) | 72.60 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity and race identities overlapped for some participants (e.g., Hispanic and Black). Other participants reported their race and ethnicity as Hispanic.
  Participants
    number analyzed (Participants) | 9 | 9 | 18
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 2 | 6
    White | 3 | 5 | 8
    More than one race | 2 | 2 | 4
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Birthweight [Mean (Standard Deviation); unit: oz] | 118.33 (13.74) | 111.53 (14.86) | 114.93 (14.48)
Body Mass Index Percentile (calculated from WHO Growth Charts) [Mean (Standard Deviation); unit: percentile] | 51.69 (28.41) | 53.85 (28.95) | 52.77 (28.20)

OUTCOME MEASURES:

1. Primary Outcome: Group Differences in Infant BMI
Description: Families receiving the program will be compared to infants in control families who receive standard ECS content only to determine which group has a lower proportion of infants with Body Mass Index greater than or equal to the 85th percentile.
  Anthropometrics were measured in triplicate using a calibrated mobile digital SECA baby scale and portable infant length board. Infants were weighed in a clean diaper without clothes to the nearest 1 gram. All length measurements were performed by two team members.
  Infant BMI standardized for age and sex was calculated from the WHO 2005 growth standards to obtain BMI percentile. Percentiles under the 5th percentile are considered underweight, percentiles between 5th- 85th percentile are considered healthy weight, percentiles 85th- 95th percentile are considered overweight, and percentiles equal to or greater than the 95th percentile are considered obesity.
Time Frame: The measure of group differences in infant BMI will be completed at post-treatment (when the child is 9 months of age).
Population: Was the participants post BMI > 85th
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Eating for My Infant Intervention | Control
Number analyzed (Participants) | 14 | 13
Participants
  participants post BMI > 85th | 5 | 2
  participants post BMI < 85th | 9 | 11

2. Secondary Outcome: Group Differences in Infant Diet Quality
Description: Diet will be assessed via three random dietary recall interviews conducted with mothers by phone. Trained interviewers, blinded to participant study condition, will employ the United States Department of Agriculture (USDA) automated multiple-pass method (AMPM), a standardized interview approach. Differences between the control and intervention group on diet quality (Healthy Eating Index; HEI) at post-treatment were calculated. Scores range from 0- 100 with higher scores representing greater diet quality.
  Footnote: Originally proposed study outcomes included examination of pre-post changes in diet by treatment group (e.g., food groups) but this analysis was not possible because at baseline infants were 2 months of age and not yet consuming any solid foods.
Time Frame: The measure of infant diet will be completed within 2 weeks of the baseline visit (when the child is 2 months of age) and again within 2 weeks of the post-treatment visit (when the child is 9 months of age).
Population: Data from dietary recalls at post-treatment (age nine months) will be used to calculate diet quality using the new Healthy Eating Index (HEI-Toddlers-2020) for children under two years of age.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Eating for My Infant Intervention | Control
Number analyzed (Participants) | 14 | 14
score on a scale | 47.57 (7.20) | 46.50 (7.70)

3. Secondary Outcome: Group Differences in Infant Diet Diversity
Description: Diet will be assessed via three random dietary recall interviews conducted with mothers by phone within 2 weeks of the baseline and post-treatment study visit dates. Trained interviewers, blinded to participant study condition, will employ the United States Department of Agriculture (USDA) automated multiple-pass method (AMPM), a standardized interview approach. Differences between the control and intervention group on diet diversity (Minimum Diet Diversity) at post-treatment were calculated. Adequate MDD is defined as consuming a food from 4 or more of seven food groups in any amount during the prior 24 hours (possible score range 0- 7).
  Footnote: Originally proposed study outcomes included examination of pre-post changes in diet by treatment group (e.g., food groups) but this analysis was not possible because at baseline infants were 2 months of age and not yet consuming any solid foods.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: food groups
Arm/Group | Healthy Eating for My Infant Intervention | Control
Number analyzed (Participants) | 14 | 14
food groups | 4.24 (1.13) | 4.01 (1.13)

4. Secondary Outcome: Treatment Acceptability
Description: Family perception of program acceptability was reported using an established questionnaire assessing components of the theoretical framework of acceptability (TFA; Timm et al., 2022) with minor wording adaptations to better fit the HEMI program. The total measure included 3 subscale scores: Affective attitude and effectiveness, coherence and understanding, and perceived burden (Timm et al., 2022). A single overall acceptability question was also included. Scores were scaled to 100 with a score of 100 representing highest acceptability and 20 representing the lowest acceptability.
Time Frame: The measure of feedback on the intervention will be completed at post-treatment (when the child is 9 months of age).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Eating for My Infant Intervention
Number analyzed (Participants) | 13
units on a scale
  Overall Acceptability | 94.29 (9.38)
  Affective attitude and effectiveness | 89.17 (8.72)
  Coherence and understanding | 88.10 (10.52)
  Perceived burden | 65.00 (18.29)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the intervention period and at post-treatment assessment (6 months).
Description: Mild: An event that is easily tolerated by the subject, causing minimal discomfort and not interfering with everyday activities. Moderate: An event that is sufficiently discomforting to interfere with normal everyday activities. Severe: An event that prevents normal everyday activities. AEs were collected at each intervention session (Session 1, Session 2, Session 4, Session 5) and at post treatment for both intervention and control families.
Arm/Group | Healthy Eating for My Infant Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 5/15 | 4/15
Other Adverse Events (participants affected / at risk) | 14/15 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Eating for My Infant Intervention (N=15) | Control (N=15)
RSV (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Ear Infection (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Flu/Virus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Swollen Nodes (Immune system disorders) | 0 (0) | 1 (1)
Flu/Virus (Immune system disorders) | 1 (1) | 1 (1)
NJ/NG Tube Surgery (Surgical and medical procedures) | 0 (0) | 1 (2)
Croup (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Eating for My Infant Intervention (N=15) | Control (N=15)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3)
Allergic Reaction (Immune system disorders) | 1 (3) | 2 (3) — swollen, rash, hives,
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eye Irritation (Eye disorders) | 1 (1) | 1 (1) — pinkeye, eye mucus
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Surgical Procedure (Surgical and medical procedures) | 3 (3) | 1 (1) — circumcision, surgical removal of growth on foot
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) — child fell
Hearing Difficulties (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Acid Reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (3)
Ear Infection (Ear and labyrinth disorders) | 3 (3) | 3 (3)
Fever (Immune system disorders) | 4 (5) | 0 (0)
Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Viral Infections (Immune system disorders) | 3 (3) | 4 (6) — RSV, COVID-19, cold, flu, virus, upper respiratory

LIMITATIONS AND CAVEATS:
This study used a small sample size, limiting power for identifying efficacy. Given the small sample, we were unable to conduct an analysis to identify the benefit of each component. Given families were allowed to select modules, each family received a different combination of modules. Different modules may have had varied impact on study outcomes; our study was unable to explore the impact of individual modules or variations of combinations of modules.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT04977947/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT04977947/SAP_001.pdf
  • Informed Consent Form (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT04977947/ICF_002.pdf